CLINICAL TRIAL: NCT06762275
Title: Optimizing Management of Children Presenting With Acute Abdominal Pain in Primary Care: a Cluster Randomized Controlled Trial Evaluating the Impact of a Clinical Prediction Rule Including C-reactive Protein for Appendicitis
Brief Title: The Impact of a Diagnostic Strategy for Acute Appendicitis in Children With Acute Abdominal Pain in Primary Care
Acronym: ISAAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Leiden University Medical Center (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: METc 2022/399; 10390022210064 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2024-12-03; First posted 2025-01-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Appendicitis Acute; Acute Abdomen in Children
Keywords: General practitioner; Appendicitis; Clinical prediction rule; C-reactive protein; Children
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Even though the GP's and children can not be blinded to the allocation, researchers performing the analyses will be blinded to the assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnostic strategy (Experimental): GPs in the intervention group will use a diagnostic strategy for AA referral, consisting of an externally validated cPR based on seven signs and symptoms, selectively followed by CRP-POCT in children in the medium risk group according to the cPR.
  Interventions: Diagnostic Test: Diagnostic strategy
- Control (No Intervention): GPs in the control group provide care as usual, i.e. according to the Dutch College of GPs (NHG) guideline 'Abdominal pain in children', which does not include specific recommendations for AA referral and in which CRP POCT is not recommended. See for details: Detailed description - Usual care.

INTERVENTIONS:
Diagnostic Test: Diagnostic strategy — GPs' use of an externally validated cPR followed by CRP-POCT in the medium risk group. See for details: Detailed description - Intervention.
  Other Names: Clinical prediction rule; C-reactive protein point-of-care test
  Arms: Diagnostic strategy

SUMMARY:
BACKGROUND Acute appendicitis (AA) in an early stage is difficult to distinguish from other (self-limiting) causes of acute abdominal pain (e.g. constipation and gastroenteritis), resulting in missing 19% of children with AA at first presentation in primary care and 70% of non-AA cases among referrals.

OBJECTIVE To evaluate the impact of the use of a diagnostic strategy for acute appendicitis (AA), which consists of a clinical prediction rule (cPR) including C-reactive protein point-of-care test (CRP POCT), on referral efficiency in children with acute abdominal pain in primary care, as compared to usual care.

STUDY DESIGN This is a cluster randomized controlled trial in primary care with a process evaluation. GPs in the intervention group will use an externally validated cPR based on symptoms and signs selectively followed by a CRP POCT in the medium risk group. GPs from general practices allocated to the control group will provide care and diagnosis as usual, i.e. following recommendations of the Dutch College of GPs guideline 'abdominal pain in children'.

STUDY POPULATION Children aged 4 to 18 years presenting to their general practitioner (GP) with acute abdominal pain.

OUTCOME MEASURES Primary outcome: referral efficiency (proportion non-referrals in non-AA patients during 30 days follow-up).

Secondary outcomes: safety (proportion of referrals in AA patients during the first consultation), proportion of children with CRP-POCT, proportion of children with planned reassessment, child anxiety, parent or child satisfaction, quality of life, and costs.

DETAILED DESCRIPTION:
BACKGROUND About 10% of pediatric general practitioner (GP) consultations are for acute abdominal pain of which about 5% have acute appendicitis (AA). Delaying a diagnosis of AA and subsequent appendectomy increases the short and long-term morbidity. AA in an early stage is difficult to distinguish from other (self-limiting) causes of acute abdominal pain (e.g. urinary tract infection, constipation and gastroenteritis), resulting in missing 19% of children with AA at first presentation in primary care and 70% non-AA cases among referrals, which has a negative impact on the child and parents, such as anxiety and psychological distress.

As urgent illnesses other than AA are very rare in children with acute abdominal pain, the yield of referrals in terms of detecting other conditions than AA that need urgent specialist care is low. An evidence based diagnostic strategy for AA referral could help the GP in the diagnostic process, thereby reducing non-AA referrals without missing children with AA.

OBJECTIVE AND HYPOTHESIS The objective of this study is to evaluate the impact of a diagnostic strategy for AA, consisting of an externally validated cPR based on seven signs and symptoms, selectively followed by a CRP-POCT in the medium-risk group, on referral efficiency in children with acute abdominal pain in primary care, as compared with usual care. The hypothesis is that the diagnostic strategy will decrease the proportion of non-AA referrals, without delaying the diagnosis of AA.

STUDY DESIGN A pragmatic cluster RCT will be conducted with 1:1 permuted-block randomization of general practices to the intervention or control group using randomly varying block size. Stratification will be based on the GP practice size (greater or smaller than 5000 patients). Follow-up is 30 days for the primary outcome (efficiency) and 30 days and 3 months for secondary outcomes (7). Alongside the trial, a process evaluation will be performed according to the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance).

STUDY POPULATION Inclusion criteria are: children, 4 to 18 years, presenting with acute abdominal pain (onset ≤ 7 days) in primary care.

Exclusion criteria are: a history of appendectomy, pregnancy, traumatic cause of abdominal pain.

INTERVENTION The intervention in this study is a diagnostic strategy for AA referral using an externally validated cPR selectively followed by a CRP POCT in the medium risk group. By using the diagnostic strategy, GPs will evaluate a set of signs and symptoms on a structural basis and get guidance for indication and interpretation of CRP POCT, for which current practice is very heterogeneous. The cPR includes seven signs and symptoms of AA: sex (2 points), duration of symptoms (< 24 hrs= 1 point, 24-48 hrs= 2 points), nausea or vomiting (2 points), elevated temperature (≥ 37.3 °C) (1 point), tenderness of the right lower quadrant (5 points), peritoneal irritation (4 points), and abnormal bowel sounds (1 point). For children in the low-risk group (score 0-7; mean probability AA 0.5%) safety netting advice should be provided. In the high-risk group (score ≥14; mean probability AA 41.0%), the GP should refer the patient to the emergency department. In the medium-risk group (score 8-13; mean probability AA 7.5%), GPs should perform CRP POCT according to Dutch laboratory quality standards. CRP values <10mg/l (mean probability AA 1.3%) imply safety netting advice and for CRP >50 mg/l a referral is needed (mean probability AA 41.8%). In case of a CRP value between 10 and 50 mg/l (mean probability AA 16.8%), the GP will discuss the following two management options with the patient: 1) a reconsultation later the same day or the next day; or 2) immediate referral. The cPR will be made available electronically for GPs, by a link integrated in the GP registry.

USUAL CARE Care provided as usual is according to the recommendations of the Dutch College of GPs guideline 'abdominal pain in children', which states that AA could be suspected when a child presents with pain and tenderness in the right lower quadrant and fever. Children with peritonitis signs and abnormal bowel sounds need to be referred. In case of doubt, GPs should perform safety netting and/or plan reassessment. CRP testing is not recommended, because lack of evidence for added diagnostic value in primary care. The GPs in the control group receive a leaflet with a summary of the NHG guideline 'abdominal pain in children'.

SAMPLE SIZE CALCULATION Results from previous studies show that the cut-off for the high-risk group based on the cPR had a specificity of 97% and that CRP value of ≥50 mg/l in children in the medium risk group had a specificity of 94%. As the weighted mean of these is a specificity (efficiency) of at least 95%, an improvement of efficiency from 88% (current care) to 95% is expected. In order to detect this difference, with 80% power, using a two-sided 5% significance level, and expecting 10% loss to follow-up, a randomized controlled trial would need to include 566 children (283 per group). The researchers assume to recruit on average 4 children per practice in 2 years and that 10 practices will not recruit any children. Therefore, 150 practices will be recruited which each recruit children for 2 years.

STATISTICAL ANALYSIS The primary outcome will be evaluated on an intention-to-treat basis. Children will be analyzed in the intervention or control group based on the GP practice in which they are registered, irrespective of the actual care received. In addition, a per protocol analysis will be done. In the intervention group according to the per protocol analysis, only children who received the intended diagnostic strategy and CRP-POCT testing in the prescribed way will be included. In the control group, we will only include children who did not undergo CRP POCT testing. Separately in both randomized groups, characteristics of children will be compared in the intention-to-treat and per-protocol analysis. A multilevel logistic regression model will be used to analyze the primary outcome, accounting for clustering of observations within GP practices and adjusting for the stratification variable (practice size) and, if necessary, for baseline differences. Exploratory analyses will assess subgroups by age and sex.

For secondary outcomes, multilevel logistic (dichotomous variables) or linear regression (continuous variables) will be used, as appropriate. In addition, adverse health outcomes (e.g. complications in AA cases and non-AA cases, missed other emergency diseases) will be described without statistical evaluation.

COST-EFFECTIVENESS ANALYSIS Cost-effectiveness will be calculated from societal and healthcare perspective with a time horizon of 30 days. Secondary analyses will address a 3-month time horizon. Efficiency will be the primary effect parameter. Cost-utility will be calculated based on the EQ-5D-(Y)-3L. Bootstrap re-sampling will be performed on the costs, and on costs and effect pairs (cost-effectiveness and cost-utility analyses) in order to calculate confidence intervals. Furthermore, both cost-effectiveness and cost-utility planes will be plotted, along with acceptability curves.

ELIGIBILITY:
Inclusion criteria:

- Children aged 4 to 18 years with acute abdominal pain (onset ≤ 7 days) who present at the GP.

Exclusion criteria:

* A history of appendectomy
* Current pregnancy
* Traumatic cause of abdominal pain

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 566 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Referral efficiency | 30 days follow-up from baseline
  The referral efficiency is defined as the proportion of non-referrals in patients without AA during 30 days follow-up (development of appendicitis beyond this period is extremely unlikely). This corresponds with the specificity of the diagnostic strategy. Medical records of the participating children in the GPs registry, including discharge letters (hospital data), will be screened by the researchers, in order to assess whether children were referred and whether they were or were not diagnosed with AA.

SECONDARY OUTCOMES:
Safety | 30 days follow-up from baseline
  The safety is defined as the proportion of referrals in patients with AA during first consultation at the GP (baseline). This corresponds with the sensitivity of the diagnostic strategy. Medical records of the participating children in the GPs registry, including discharge letters (hospital data), will be screened by the researchers, in order to assess whether children were referred and whether they were or were not diagnosed with AA.
Proportion of children with CRP-POCT | Baseline
  Proportion of children with a CRP-POCT in primary care among all children per randomized group at baseline. The researchers will review data from the GP registry to identify whether a CRP-POCT was carried out for each child.
Proportion of children with planned reassessment | Baseline
  Proportion of children with planned reassessment in all children per randomized group at baseline. The researchers will use GP registry data to determine whether a reassessment was planned for each child. GPs will be explicitly instructed to document in the medical files whether a reassessment was planned or unplanned.
Anxiety of child ≥8 years according to the Dutch version of the State-Trait Anxiety Inventory for Children | 30 days and 3 months follow-up from baseline
  Children ≥8 years will complete the Dutch version of the State-Trait Anxiety Inventory for Children (STAIC) questionnaire. It measures self-perceived anxiety in children based on two scales: state-anxiety and trait-anxiety. The Dutch version of the STAIC (Zelfbeoordelingsvragenlijst voor Kinderen (ZBV-K) Versie Nu) questionnaire consists only of the state-anxiety scale. The questionnaire consists of 20 statements involving the current state of mind of the child. The score ranges from 20 to 60. The higher the score, the higher the level of state-anxiety of the child.
Parent or child satisfaction with management according to the Parental Medical Interview Scale (P-MISS) | 30 days follow-up from baseline
  Parents (for children 4-15 years) or children (16-18 years) will complete a Dutch translation of the P-MISS questionnaire. This questionnaire is used to measure the satisfaction of parents or children with the consultation at their GP for acute abdominal pain. The questionnaire consists of 26 statements about different aspects of the consultation. The child or parent has to rank each statement based on a Likert scale (1= do not agree at all, 5= totally agree). The maximum score is 130 and the minimum score is 26. The higher the score, the higher the satisfaction level.
Quality of life of child according to the EuroQol 5D (EQ-5D) | 30 days and 3 months follow-up from baseline
  For children ≤7 years, parents will complete the proxy version of the EQ-5D-3L. Children 8-15 years will complete the EQ-5D-youth and children ≥16 years will complete the EQ-5D questionnaire. The EQ-5D-3L is a standardized instrument which assesses the health-related quality of life of the child based on five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (0), some problems (1), and extreme problems (2). The maximum score is 10 and the minimal score is 0. The EQ VAS records the parent- or self-rated current health of the child on a vertical analogue scale ranging from 0 ('Worst' to 100 ('Best').
Costs (societal and healthcare perspective) | 30 days and 3 months follow-up from baseline
  The costs for the effectiveness analysis and cost-utility analysis will be based upon an adapted version of the iMTA Productivity Costs Questionnaire (iPCQ) and iMTA Medical Consumption Questionnaire (iMCQ), through which data on health care consumption and productivity losses will be collected. Parents (for children ≤15 years) and/or children (≥16 years) will complete the adapted version of these questionnaires, which consists of a total of 16, respectively 18, questions about healthcare consumption, costs and productivity losses caused by abdominal complaints of the child. The units measured (medical consumption and productivity losses) will be monetarized according to guidelines of the National Healthcare Institute of the Netherlands. Thereafter, the costs of all items will be summed and weighted in conjunction with the outcomes in order to inform policymakers.

CONTACTS AND LOCATIONS:
Overall Officials: Gea A. Holtman, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Processed and pseudonymized data, syntaxes, data documentation and raw data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After all publications concerning the study are published.
Access Criteria: Data will be made available upon reasonable request. In addition, processed and pseudonymized data will be made available upon restricted access (DataverseNL). Meta data will be presented in the UMCG Research Data Catalogue. DOI (Digital Object Identifier) will be shared via publications to make the data more findable.

REFERENCES:
- [Background] Blok GCGH, Veenstra LMM, van der Lei J, Berger MY, Holtman GA. Appendicitis in children with acute abdominal pain in primary care, a retrospective cohort study. Fam Pract. 2021 Nov 24;38(6):758-765. doi: 10.1093/fampra/cmab039. PMID 34278425
- [Background] Gorter RR, Eker HH, Gorter-Stam MA, Abis GS, Acharya A, Ankersmit M, Antoniou SA, Arolfo S, Babic B, Boni L, Bruntink M, van Dam DA, Defoort B, Deijen CL, DeLacy FB, Go PM, Harmsen AM, van den Helder RS, Iordache F, Ket JC, Muysoms FE, Ozmen MM, Papoulas M, Rhodes M, Straatman J, Tenhagen M, Turrado V, Vereczkei A, Vilallonga R, Deelder JD, Bonjer J. Diagnosis and management of acute appendicitis. EAES consensus development conference 2015. Surg Endosc. 2016 Nov;30(11):4668-4690. doi: 10.1007/s00464-016-5245-7. Epub 2016 Sep 22. PMID 27660247
- [Background] Blok G, Burger H, van der Lei J, Berger M, Holtman G. Development and validation of a clinical prediction rule for acute appendicitis in children in primary care. Eur J Gen Pract. 2023 Dec;29(1):2233053. doi: 10.1080/13814788.2023.2233053. PMID 37578416
- [Background] Blok GCGH, Nikkels ED, van der Lei J, Berger MY, Holtman GA. Added value of CRP to clinical features when assessing appendicitis in children. Eur J Gen Pract. 2022 Dec;28(1):95-101. doi: 10.1080/13814788.2022.2067142. PMID 35535699
- [Background] Kharbanda AB, Vazquez-Benitez G, Ballard DW, Vinson DR, Chettipally UK, Dehmer SP, Ekstrom H, Rauchwerger AS, McMichael B, Cotton DM, Kene MV, Simon LE, Zhu J, Warton EM, O'Connor PJ, Kharbanda EO; Clinical Research on Emergency Services and Treatments Network (CREST) and the Critical Care Research Center, HealthPartners Institute. Effect of Clinical Decision Support on Diagnostic Imaging for Pediatric Appendicitis: A Cluster Randomized Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2036344. doi: 10.1001/jamanetworkopen.2020.36344. PMID 33560426
- [Background] Lintula H, Kokki H, Kettunen R, Eskelinen M. Appendicitis score for children with suspected appendicitis. A randomized clinical trial. Langenbecks Arch Surg. 2009 Nov;394(6):999-1004. doi: 10.1007/s00423-008-0425-0. Epub 2008 Oct 8. PMID 18841382
- [Background] Ansems S, Berger M, Rheenen PV, Vermeulen K, Beugel G, Couwenberg M, Holtman G. Effect of faecal calprotectin testing on referrals for children with chronic gastrointestinal symptoms in primary care: study protocol for a cluster randomised controlled trial. BMJ Open. 2021 Jul 23;11(7):e045444. doi: 10.1136/bmjopen-2020-045444. PMID 34301652
- [Background] Kappen TH, van Loon K, Kappen MA, van Wolfswinkel L, Vergouwe Y, van Klei WA, Moons KG, Kalkman CJ. Barriers and facilitators perceived by physicians when using prediction models in practice. J Clin Epidemiol. 2016 Feb;70:136-45. doi: 10.1016/j.jclinepi.2015.09.008. Epub 2015 Sep 21. PMID 26399905
- [Background] van der Wouden JC, Blankenstein AH, Huibers MJ, van der Windt DA, Stalman WA, Verhagen AP. Survey among 78 studies showed that Lasagna's law holds in Dutch primary care research. J Clin Epidemiol. 2007 Aug;60(8):819-24. doi: 10.1016/j.jclinepi.2006.11.010. Epub 2007 Mar 26. PMID 17606178
- [Background] Bjarnason NH, Kampmann JP. Selection bias introduced by the informed consent process. Lancet. 2003 Jun 7;361(9373):1990. doi: 10.1016/S0140-6736(03)13568-4. No abstract available. PMID 12801770
- [Background] Van den Bruel A, Jones C, Thompson M, Mant D. C-reactive protein point-of-care testing in acutely ill children: a mixed methods study in primary care. Arch Dis Child. 2016 Apr;101(4):382-5. doi: 10.1136/archdischild-2015-309228. Epub 2016 Jan 12. PMID 26757989
- [Background] Adams G, Gulliford MC, Ukoumunne OC, Eldridge S, Chinn S, Campbell MJ. Patterns of intra-cluster correlation from primary care research to inform study design and analysis. J Clin Epidemiol. 2004 Aug;57(8):785-94. doi: 10.1016/j.jclinepi.2003.12.013. PMID 15485730
- [Background] Schols AM, Dinant GJ, Cals JW. Point-of-care testing in general practice: just what the doctor ordered? Br J Gen Pract. 2018 Aug;68(673):362-363. doi: 10.3399/bjgp18X698033. No abstract available. PMID 30049755
- [Background] Schunemann HJ, Oxman AD, Brozek J, Glasziou P, Jaeschke R, Vist GE, Williams JW Jr, Kunz R, Craig J, Montori VM, Bossuyt P, Guyatt GH; GRADE Working Group. Grading quality of evidence and strength of recommendations for diagnostic tests and strategies. BMJ. 2008 May 17;336(7653):1106-10. doi: 10.1136/bmj.39500.677199.AE. PMID 18483053
- [Background] RIFT Study Group on behalf of the West Midlands Research Collaborative. Appendicitis risk prediction models in children presenting with right iliac fossa pain (RIFT study): a prospective, multicentre validation study. Lancet Child Adolesc Health. 2020 Apr;4(4):271-280. doi: 10.1016/S2352-4642(20)30006-7. Epub 2020 Feb 13. PMID 32200936